CLINICAL TRIAL: NCT03317912
Title: Effect of Peroperative Intravenous Infusion of Lignocaine on the Quality of Postoperative Sleep
Brief Title: Perioperative Lignocaine and Sleep Disturbance
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Jean François Brichant, Professor, University of Liege
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ULiege
Record Dates: First submitted 2015-03-31; First posted 2017-10-23 (Actual); Last update posted 2017-10-23 (Actual); Status verified 2017-10

CONDITIONS: Sleep Disturbance
MeSH Terms: conditions — Parasomnias | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lidocaïne 2% (Active Comparator): Bolus 0.075ml/kg/h, following by continuous infusion 0.1ml/kg/h during surgery and 0.066ml/kg/h during 24h
  Interventions: Drug: Lidocaïne 2%
- Placebo (for Lidocaïne) (Placebo Comparator): Bolus 0.075ml/kg/h, following by continuous infusion 0.1ml/kg/h during surgery and 0.066ml/kg/h during 24h
  Interventions: Drug: Placebo (for Lidocaïne)

INTERVENTIONS:
Drug: Lidocaïne 2% — Continuous infusion during per and postoperative periods
  Other Names: lignocaïne; Linisol
  Arms: Lidocaïne 2%
Drug: Placebo (for Lidocaïne) — Continuous infusion during per and postoperative periods
  Other Names: NaCl 0.9%
  Arms: Placebo (for Lidocaïne)

SUMMARY:
The aim of this clinical trial is to study the effect of an intravenous infusion of lidocaïne in a multimodal analgesic protocol on the architecture sleep during the first postoperative night.

DETAILED DESCRIPTION:
To study the effect of lidocaïne, we plan to include 40 patients, randomized in 2 groups, undergoing open prostate surgery in this randomized placebo-controlled trial.

Before anesthesia induction, these patients receive an intravenous lidocaine infusion (bolus 1,5 mg.kg-1 followed by a continuous infusion of 2mg.kg-1.h during 24 hours) or an equal volume of placebo. Then the anesthesia is induced with propofol, sufentanil et rocuronium. The postoperative analgesia is provided by paracetamol, tramadol and patient-controlled analgesia (PCA) with morphine or oral oxycodone. A polysomnography is registred on the preoperative night and on the first postoperative night.

ELIGIBILITY:
Inclusion Criteria:

* Radical prostatectomy

Exclusion Criteria:

* BMI > 30
* Neurologic/psychiatric diseases or therapeutics, seizyres
* Cardiac disease, second or third degree atrioventricular block
* Obstructive sleep apnea syndrome
* History of liver or renal insufficiency
* and any contraindication to the anesthetic protocol of the study.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-12 (Estimated); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Time ratio between rapid eye movement sleep(REM) + Stage 3 sleep / Stage 1 + Stage 2 sleep | Postoperaty day 1

SECONDARY OUTCOMES:
Sleep latence | Postoperaty day 1
Sleep time | Postoperaty day 1
Cumulative Opioid use | Postoperaty day 1
Quality of analgesia (Visual Analogic Scale) | Postoperaty day 1

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Maquoi, Principal Investigator — CHU Liege - Department of Anesthesia and Intensive Care Medicine

REFERENCES:
- [Result] Kaba A, Laurent SR, Detroz BJ, Sessler DI, Durieux ME, Lamy ML, Joris JL. Intravenous lidocaine infusion facilitates acute rehabilitation after laparoscopic colectomy. Anesthesiology. 2007 Jan;106(1):11-8; discussion 5-6. doi: 10.1097/00000542-200701000-00007. PMID 17197840
- [Result] Krenk L, Jennum P, Kehlet H. Postoperative sleep disturbances after zolpidem treatment in fast-track hip and knee replacement. J Clin Sleep Med. 2014 Mar 15;10(3):321-6. doi: 10.5664/jcsm.3540. PMID 24634631